CLINICAL TRIAL: NCT00508443
Title: Phase I/II Evaluation of a Novel CT-On-Rails or Trilogy Stereotactic Spine Radiotherapy System (SSRS) for the Treatment of Metastatic Spine Disease
Brief Title: Evaluation of a Novel CT-On-Rails or Trilogy Stereotactic Spine Radiotherapy System (SSRS)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-446; NCI-2012-01584 (Registry Identifier: NCI CTRP); ID02-446 (Other: MD Anderson)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Spinal Neoplasms
Keywords: Stereotactic Spine Radiotherapy System; SSRS; CT-on-Rails; Metastatic Spine Disease; Spinal Neoplasms; Radiation Therapy; Trilogy; Cancer; Breast Cancer; Gastrointestinal Cancer; Genitourinary Disease; Lung Cancer; Lymphoma; Melanoma; Sarcoma; Spinal Cancer
MeSH Terms: conditions — Spinal Neoplasms; Spinal Diseases; Neoplasms; Breast Neoplasms; Gastrointestinal Neoplasms; Urogenital Diseases; Lung Neoplasms; Lymphoma; Melanoma; Sarcoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation Therapy (Experimental): Radiation Therapy using CT-on-Rails or Trilogy procedure. Participants prescribed to receive 9 Gy x 3 so that a peripheral dose of 27 Gy is given to the tumor.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Three radiation treatments guided by the CT-on-Rails or Trilogy procedure over a period of 2 weeks. Participants prescribed to receive 9 Gy x 3 so that a peripheral dose of 27 Gy is given to the tumor.

SUMMARY:
The goal of this clinical research study is to find out if stereotactic spine radiotherapy is safe and effective in the treatment of metastatic spine tumors. The feasibility of this type of treatment will be studied as will any side effects related to the treatment. The precision and accuracy of the CT-on-rails will also be studied.

DETAILED DESCRIPTION:
CT-On-Rails or Trilogy is a system that places the radiation treatment machine in the same room as the CT scanner so that the CT scanner can help deliver radiation more precisely.

You will have a MRI of the spine within 1 month of registration on this study. You will also fill out a health survey (5 minutes), a symptom inventory ( 5 minutes), and a Brief Pain Inventory (5 minutes) within 1 week of registration.

A pretreatment feasibility study will first be performed to determine the precision, accuracy, and reproducibility with which the target volume and critical normal structures (e.g. spinal cord) can be positioned relative to the radiation beams for spine tumors; this will consist of a CT scan.

Patients will have a CT-simulation. The simulation is like a CT scan where a special body frame is used to keep the patient from moving during scanning and later treatment.

You will be asked questions about your medical history and have a complete neurological exam during your first consultation. The neurological exam involves testing upper and lower motor strength, sensation to light touch, reflexes, mental exam, and way you walk. MRI of the spine must be performed within 1 month of registration. You will be asked to complete 3 questionnaires to evaluate your symptoms and pain. Each questionnaire will take around 5 minutes to complete, and should be completed within 1 month of being enrolled in the study.

All patients will be treated with radiation therapy that is guided by the CT-on-Rails or Trilogy procedure. Patients will receive a CT scan immediately before the treatment in the same room of the treatment using CT-On-Rails or Trilogy. There will be a total of 3 treatments over a period of 2 weeks.

Monitoring of side effects will be focused on neurological, gastrointestinal, musculoskeletal, and hematological systems. Every attempt will be made to have the patient complete the prescribed course of radiation to maximize the beneficial effect of treatment. However, if there is severe side effects, radiation treatment will be stopped and patients will be taken off study.

You will have follow up visits once a week during radiation treatment, scheduled on the same day as radiation. After treatment, you will have telephone, mail, or follow-ups per fax scheduled at 2 and 4 weeks,and 2 months post radiation. You will have follow up visits scheduled at 3, 6, 9, 12, 18, and 24 months, then every six months for the rest of your life. At all follow-up visits, you will be asked questions about your medical history, have a neurological exam, and neurologic function will be evaluated. Any pain medication you are taking will be noted. You will have an MRI of the spine at 3, 6, 9, 12,18, and 24 months, then once a year for the rest of your life. You will also be asked to complete 3 questionnaires to evaluate your symptoms and pain. Each questionnaire will take around 5 minutes to complete.

This is an investigational study. The CT-on-rails and Trilogy linear accelerator are FDA-approved medical devices and are commercially available, however, the way these two devices are being used is investigational. Up to 150 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographically documented spine or paraspinal metastasis demonstrated on spine MRI within 4 wks of registration
2. Maximum of 2 metastatic sites in the spine to be irradiated over a single course of treatment.
3. Informed consent for irradiation or re-irradiation of spinal or para-spinal tumor (s)
4. Diagnosis cancer including but not limited to lung (non-small cell and small cell), breast, prostate, renal cell, melanoma, gastrointestinal, germ cell tumors, and unknown primary tumors
5. Karnofsky performance status of at least 40 (i.e. not requiring active hospitalization)
6. Maximum of 1 prior course of spine radiotherapy to the current region of interest allowed.

Exclusion Criteria:

1. Worsening neurological status due to radiographic evidence of spinal cord compression requiring immediate surgical decompression or emergent conventional external radiation therapy
2. Delay in initiation of radiation treatment would be potentially detrimental to neurological outcome
3. Patients already re-treated with radiation as part of this protocol will not be eligible for additional re-treatment
4. Unstable spine requiring surgical stabilization.
5. Sites outside the spine (eg. lung, liver) are not eligible for treatment
6. Systemic radiotherapy (Sr-89) within 30 days
7. Prior irradiation of the area to be treated within 3 months of registration
8. Patients currently receiving, or who have received chemotherapy within 30 days are not eligible
9. Inability to tolerate lying flat on treatment couch for greater than 30 minutes.
10. Patient with multiple myeloma
11. Patients unable to undergo MRI of the spine
12. Patients with pacemakers
13. Patients who have previously received maximum cord tolerance of 45 Gy in 5 weeks conventional fractionation or equivalent dose to the current area to be treated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2002-10-25 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient Response (Pain Relief) | Baseline, 3, 6, 9, 12, 18, and 24 months, then every six months
  The validated Brief Pain Inventory (BPI), MD Anderson Symptom Inventory (MDASI), and SF-12v2 Health Survey used to assess changes in these indicators compared to pre-treatment baseline. Response determined by follow-up questionaires. Time to maximal pain relief is the time from the first day of irradiation until the lowest pain score for average pain after radiotherapy. The "worst pain score" from BPI used as the marker for treatment success or failure.

CONTACTS AND LOCATIONS:
Overall Officials: Amol J. Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang XS, Rhines LD, Shiu AS, Yang JN, Selek U, Gning I, Liu P, Allen PK, Azeem SS, Brown PD, Sharp HJ, Weksberg DC, Cleeland CS, Chang EL. Stereotactic body radiation therapy for management of spinal metastases in patients without spinal cord compression: a phase 1-2 trial. Lancet Oncol. 2012 Apr;13(4):395-402. doi: 10.1016/S1470-2045(11)70384-9. Epub 2012 Jan 27. PMID 22285199
- [Derived] Boehling NS, Grosshans DR, Allen PK, McAleer MF, Burton AW, Azeem S, Rhines LD, Chang EL. Vertebral compression fracture risk after stereotactic body radiotherapy for spinal metastases. J Neurosurg Spine. 2012 Apr;16(4):379-86. doi: 10.3171/2011.11.SPINE116. Epub 2012 Jan 6. PMID 22225488
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org